CLINICAL TRIAL: NCT02433457
Title: An Open-label, Phase 1, Randomized, Seven-treatment, Seven-period, Crossover Study to Assess the Relative Bioavailability, pH Effect, Food Effect and Dose Proportionality of CC-292 Spray Dried Dispersion Formulation in Healthy Volunteers
Brief Title: Relative Bioavailability Study of CC-292
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-292-CP-002
Record Dates: First submitted 2015-03-26; First posted 2015-05-05 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; CC-292; Open-Label; Bioavailability Pharmacokinetics; Phase I
MeSH Terms: interventions — spebrutinib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- CC-292 SDD (Spray Dried Dispersion)300mg - Fasted Condition (Experimental): Single oral dose of 300 mg CC-292 SDD under fasted conditions (100 mg SDD x 3 tablets)
  Interventions: Drug: CC-292
- CC-292 SDD 300mg - Fed Condition (Experimental): Single oral dose of 300 mg CC-292 SDD under fed conditions (100 mg SDD x 3 tablets)
  Interventions: Drug: CC-292
- 375mg P22 - Fasted condition (Experimental): Single oral dose of 375 mg P22 under fasted conditions (125 mg P22 x 3)
  Interventions: Drug: CC-292
- 375mg P22 Fed Condition (Experimental): Single oral dose of 375 mg P22 under fed conditions (125 mg P22 x 3)
  Interventions: Drug: CC-292
- CC-292 SDD 100 mg Fasted Condition (Experimental): Single oral dose of 100 mg CC-292 SDD under fasted conditions
  Interventions: Drug: CC-292
- SDD plus OMP (Oral Omeprazole) (Experimental): Single oral dose of 300 mg CC-292 SDD under fasted conditions (100 mg SDD x 3 tablets) in the presence of 40 mg
  Interventions: Drug: CC-292; Drug: Oral Omeprazole (OMP)
- P22 plus OMP (Experimental): Single oral dose of 375 mg P22 under fasted conditions (125 mg P22 x 3) in the presence of 40 mg oral OMP
  Interventions: Drug: CC-292; Drug: Oral Omeprazole (OMP)

INTERVENTIONS:
Drug: CC-292
Drug: Oral Omeprazole (OMP)
  Arms: P22 plus OMP; SDD plus OMP (Oral Omeprazole)

SUMMARY:
To evaluate the PK profile of the newly developed CC-292 SDD formulation compared to CC-292 P22 tablet.

DETAILED DESCRIPTION:
This is a single center, open-label, randomized, seven-treatment, seven-period, crossover design. The study will consist of a screening phase, a treatment phase, and a follow-up phone call. Approximately 24 healthy adult subjects (male or female) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign a written Informed Consent Form (ICF) prior to any study-related assessments/procedures being conducted.
2. Must be able to communicate with the Investigator, understand, and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Must be a male or female subject from any race between 18 to 65 years of age (inclusive) at the time of signing the ICF, and in good health as determined by Physical Examinations (PE).
4. Must comply with the following acceptable forms of contraception:

   1. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception with male condoms NOT made out of natural animal membrane (e.g., latex or polyurethane condoms are acceptable) while on study drug, and for at least 90 days after the last dose of study drug.
   2. Females of childbearing potential (FCBP) 1 must have a negative pregnancy test at Screening and at Baseline (i.e., on Day -1). FCBP who engage in activity in which conception is possible must agree to use one of the following forms of contraception during their entire participation in the study and for at least 30 days after administration of the last dose of study drug:

      * Option 1: Any one of the following: non-oral hormonal contraception (e.g., injection, implant, transdermal patch, vaginal ring); intrauterine device; tubal ligation; or a partner with a vasectomy; OR
      * Option 2: Oral contraceptive pills PLUS one additional barrier method of the following: (a) male or female condom NOT made out of natural animal membrane (e.g., latex or polyurethane is acceptable); (b) diaphragm with spermicide; (c) cervical cap with spermicide; or (d) contraceptive sponge with spermicide; OR
      * Option 3: TWO of the following barrier methods: (a) male or female condom NOT made out of natural animal membrane (e.g., latex or polyurethane is acceptable); (b) diaphragm with spermicide; (c) cervical cap with spermicide; or (d) a contraceptive sponge with spermicide.

   Note: All other females must have been surgically sterilized for at least 6 months before Screening (proper documentation required), or be postmenopausal (defined as 24 months without menses before Screening, and an estradiol level of < 30 pg/mL and a plasma Follicle Stimulating Hormone (FSH) level > 40 IU/L at Screening).
5. Must have a Body Mass Index (BMI) between 18 and 33 kg/m2 (inclusive).
6. No clinically significant laboratory test results, as determined by the Investigator.
7. Must be afebrile, with supine systolic BP of 90 to 140 mmHg, a supine diastolic Blood Pressure (BP) of 60 to 90 mmHg, and pulse rate of 40 to 110 bpm.
8. Must have a normal or clinically acceptable 12-lead Electrocardiogram (ECG) at Screening. Male subjects must have a QTcF value ≤ 430 msec. Female subjects must have a QTcF value ≤ 450 msec.

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study, or confounds the ability to interpret data from the study.
3. Use of any prescribed systemic or topical medication (including but not limited to antibiotics, analgesics, anesthetics, etc.) prior to 30 days of the first dose administration, unless Sponsor agreement is obtained.
4. Use of any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 7 days of the first dose administration, unless Sponsor agreement is obtained.
5. Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism and excretion (e.g., bariatric procedure), or plans to have elective or medical procedures during the conduct of the trial. Subjects post cholecystectomy and post appendectomy may be included.
6. Exposure to an investigational drug within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
7. Donated blood or plasma prior to 4 weeks before the first dose administration to a blood bank or blood donation center.
8. History of multiple drug allergies (i.e., two or more);
9. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) prior to 2 years before first dose administration, or a positive drug screen reflecting consumption of illicit drugs.
10. History of alcohol abuse (as defined by the current version of the DSM) prior to 2 years before dosing, or a positive alcohol screen.
11. Known to have hepatitis, or known to be a carrier of the Hepatitis B Surface Antigen (HBsAg), or Hepatitis C Virus Antibody (HCVAb), or have a positive result to the test for HBsAg, HCVAb, or Human Immunodeficiency Virus (HIV) antibodies at Screening.
12. History of smoking or the use of nicotine containing products prior to 3 months of Screening by self reporting.
13. Female subjects lactating or breastfeeding a child.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2014-09-26 (Actual); Study Completion 2014-09-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | 48 hours
  Maximum observed concentration in plasma
Pharmacokinetics - AUC 0-t | 48 hours
  Area under the plasma concentration-time curve from time zero to the last measured time point
Pharmacokinetics - AUC 0-24 | 48 hours
  Area under the plasma concentration-time curve to 24 hours post dose
Pharmacokinetics - AUC 0-∞ | 48 hours
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - %AUCextrap | 48 hours
  Percent Area under the plasma concentration-time curve extrapolated
Pharmacokinetics - Frel | 48 hours
  Relative bioavailability of the CC-292 SDD formulation compared to the reference P22 formulation
Pharmacokinetics - Tmax | 48 hours
  Time to Cmax
Pharmacokinetics - λz | 48 hours
  Terminal disposition rate constant
Pharmacokinetics - t1/2 | 48 hours
  Terminal half-life
Pharmacokinetics - CL/F | 48 hours
  Apparent clearance
Pharmacokinetics - Vz/F | 48 hours
  Apparent volume of distribution

SECONDARY OUTCOMES:
Adverse Events (AEs) | Approximatly 52 days
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Study Director — Celgene Corporation
Locations (1):
- Covance Clinical Research unit, Evansville, Indiana, United States

REFERENCES:
- [Derived] Cheng Y, Liu L, Xue Y, Zhou S, Li Y. An Open Label, Phase 1, Randomized, Seven-treatment, Seven-period, Crossover Study to Assess the Relative Bioavailability, pH Effect, Food Effect, and Dose Proportionality of CC-292, a Potent and Orally Available Bruton's Tyrosine Kinase Inhibitor. Eur J Drug Metab Pharmacokinet. 2022 Jul;47(4):579-592. doi: 10.1007/s13318-022-00776-7. Epub 2022 Jun 3. PMID 35657581